CLINICAL TRIAL: NCT02933671
Title: Suprainguinal Fascia Iliaca (SIFI) Block Improves Analgesia Following Total Hip Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving any intervention.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00070686
Record Dates: First submitted 2016-09-30; First posted 2016-10-14 (Estimated); Results first posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Hip Osteoarthritis; Primary Total Hip Arthroplasty; Pain
Keywords: suprainguinal fascia iliaca (SIFI); nerve block
MeSH Terms: conditions — Osteoarthritis, Hip; Pain | interventions — Dental Occlusion; Ropivacaine; Sodium Chloride; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suprainguinal Fascia Iliaca (SIFI) block (Experimental): A nerve block technique using a numbing medication called ropivacaine.
  Interventions: Procedure: Suprainguinal fascia iliaca (SIFI) block; Drug: Ropivacaine
- Sham group (Placebo Comparator): The same nerve block technique as above, however using an inactive solution of salt water.
  Interventions: Procedure: Sham block; Drug: Saline

INTERVENTIONS:
Procedure: Suprainguinal fascia iliaca (SIFI) block — An ultrasound guided nerve block using a medication that numbs the nerve called ropivacaine.
  Arms: Suprainguinal Fascia Iliaca (SIFI) block
Procedure: Sham block — An ultrasound guided nerve block using a medication that does NOT numb the nerve called saline, or salt water.
  Arms: Sham group
Drug: Ropivacaine — Local anesthetic (numbing drug)
  Other Names: Naropin
  Arms: Suprainguinal Fascia Iliaca (SIFI) block
Drug: Saline — Salt water placebo
  Other Names: Salt water
  Arms: Sham group

SUMMARY:
The purpose of this study is to learn if using a suprainguinal fascia iliaca (SIFI) injection technique (also called a "nerve block") that numbs the nerves going to the side and front of the upper leg will improve pain control after surgery. The SIFI technique uses a numbing solution (local anesthetics) that is injected next to nerves in the hip to reduce pain. This block may affect movement in the leg and make the legs weak. The amount of leg weakness is not known and assessment of this will be included in the study. Many institutions use the SIFI block for patients having total hip replacements, with the hope of providing good pain relief combined with improved mobility after surgery.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* between 18 and 75 years old
* American Society of Anesthesiologists (ASA) 1-3 patients undergoing primary total hip arthroplasty

Exclusion Criteria:

* ASA 4 or 5
* revision hip arthroplasty
* diagnosis of chronic pain
* daily chronic opioid use (over 3 months of continuous opioid use)
* inability to communicate pain scores or need for analgesia
* acute hip fracture
* Infection at the site of block placement
* Age under 18 years old or greater than 75 years old
* Pregnant women
* Intolerance/allergy to local anesthetics
* Weight <50 kg
* Suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, may interfere with study assessments or compliance
* Current or historical evidence of any clinically significant disease or condition that, in the opinion of the investigator, may increase the risk of surgery or complicate the subject's postoperative course.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared; patients will be deidentified and no personal information or medical records used.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suprainguinal Fascia Iliaca (SIFI) Block | Sham Group
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suprainguinal Fascia Iliaca (SIFI) Block | Sham Group | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (6.0) | 51.6 (17.8) | 57.7 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Score at 4 Hours Postoperatively, as Measured by Numerical Rating Scale (NRS) 11
Description: The NRS 11 ranges from 0 (no pain) to 10 (intense pain).
Time Frame: 4 hours postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suprainguinal Fascia Iliaca (SIFI) Block | Sham Group
Number analyzed (Participants) | 5 | 5
score on a scale | 2.4 (1.14) | 5.4 (1.95)

2. Secondary Outcome: Cumulative Opioid Consumption
Description: Reported in IV morphine equivalents.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: IV morphine equivalents in mg
Arm/Group | Suprainguinal Fascia Iliaca (SIFI) Block | Sham Group
Number analyzed (Participants) | 5 | 5
IV morphine equivalents in mg | 33.8 (24.0) | 41.9 (29.3)

3. Secondary Outcome: Motor Strength, as Measured by Dynamometry
Description: Reported as pounds per square inch (PSI).
Time Frame: 4 hours postoperatively
Measure: Mean (Standard Deviation); unit: PSI
Arm/Group | Suprainguinal Fascia Iliaca (SIFI) Block | Sham Group
Number analyzed (Participants) | 5 | 5
PSI | 28.7 (14.8) | 19.7 (22.8)

4. Secondary Outcome: Numeric Pain Score at 24 Hours, as Measured by NRS 11
Description: The NRS 11 ranges from 0 (no pain) to 10 (intense pain).
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suprainguinal Fascia Iliaca (SIFI) Block | Sham Group
Number analyzed (Participants) | 5 | 5
score on a scale | 2.6 (1.9) | 5.2 (1.3)

5. Secondary Outcome: Ambulation, as Measured by Distanced Walked
Time Frame: post-op day 0
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Suprainguinal Fascia Iliaca (SIFI) Block | Sham Group
Number analyzed (Participants) | 5 | 5
feet | 99.6 (122.2) | 20.8 (44.3)

ADVERSE EVENTS:
Time Frame: 24 hours from time of block
Arm/Group | Suprainguinal Fascia Iliaca (SIFI) Block | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Suprainguinal Fascia Iliaca (SIFI) Block (N=5) | Sham Group (N=5)
Motor weakness in the quadriceps and adductor group muscles (Musculoskeletal and connective tissue disorders) | 0 | 1 — Found to be complication of blind acetabular retractor which caused >24hr palsy in the quadriceps and adductor group muscles. Non-intervention induced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT02933671/Prot_SAP_000.pdf